CLINICAL TRIAL: NCT02203331
Title: A Randomized, Double-blind, Double-dummy, Parallel- Group, Multi-center Phase IIb Study to Assess the Efficacy and Safety of Different Dose Combinations of an Aromatase Inhibitor and a Progestin in an Intravaginal Ring Versus Placebo and Leuprorelin / Leuprolide Acetate in Women With Symptomatic Endometriosis Over a 12-week Treatment Period
Brief Title: Bay98-7196, Dose Finding / POC Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15832; 2013-005090-53 (EudraCT Number)
Record Dates: First submitted 2014-07-28; First posted 2014-07-29 (Estimated); Results first posted 2018-01-04 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Levonorgestrel; Anastrozole; Leuprolide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo (Placebo Comparator): Placebo intravaginal ring (treatment for 84 days, 28 days wearing period for each ring) and Placebo 3-months depot intramuscular injection
  Interventions: Drug: Placebo
- Levonorgestrel (Experimental): Levonorgestrel 40 µg/d intravaginal ring (treatment for 84 days, 28 days wearing period for each ring) and Placebo 3-months depot intramuscular injection
  Interventions: Drug: Placebo; Drug: Levonorgestrel
- Anastrozole 300 µg/d + Levonorgestrel (Experimental): Anastrozole 300 µg/d + Levonorgestrel 40 µg/d intravaginal ring (treatment for 84 days, 28 days wearing period for each ring) and Placebo 3-months depot intramuscular injection
  Interventions: Drug: Placebo; Drug: Anastrozole
- Anastrozole 600 µg/d + Levonorgestrel (Experimental): Anastrozole 600 µg/d + Levonorgestrel 40 µg/d intravaginal ring (treatment for 84 days, 28 days wearing period for each ring) and Placebo 3-months depot intramuscular injection
  Interventions: Drug: Placebo; Drug: Anastrozole
- Anastrozole 1050 µg/d + Levonorgestrel (Experimental): Anastrozole 1050 µg/d + Levonorgestrel 40 µg/d intravaginal ring (treatment for 84 days, 28 days wearing period for each ring) and Placebo 3-months depot intramuscular injection
  Interventions: Drug: Placebo; Drug: Anastrozole
- Lupron / Leuprolide acetate (Active Comparator): Placebo intravaginal ring (treatment for 84 days, 28 days wearing period for each ring) and Lupron / Leuprolide acetate 11.25 mg 3-months depot intramuscular injection
  Interventions: Drug: Placebo; Drug: Lupron / Leuprolide acetate

INTERVENTIONS:
Drug: Placebo — Placebo intravaginal ring (treatment for 84 days, 28 days wearing period for each ring) and Placebo 3-months depot intramuscular injection
Drug: Levonorgestrel — Levonorgestrel 40 µg/d intravaginal ring (treatment for 84 days, 28 days wearing period for each ring) and Placebo 3-months depot intramuscular injection
  Arms: Levonorgestrel
Drug: Anastrozole — Participants received Anastrozole 300 µg/d or 600 µg/d or 1050 µg/d + Levonorgestrel 40 µg/d intravaginal ring (treatment for 84 days, 28 days wearing period for each ring) and Placebo 3-months depot intramuscular injection
  Arms: Anastrozole 1050 µg/d + Levonorgestrel; Anastrozole 300 µg/d + Levonorgestrel; Anastrozole 600 µg/d + Levonorgestrel
Drug: Lupron / Leuprolide acetate — Placebo intravaginal ring (treatment for 84 days, 28 days wearing period for each ring) and Lupron / Leuprolide acetate 11.25 mg 3-months depot intramuscular injection
  Arms: Lupron / Leuprolide acetate

SUMMARY:
Purpose of the study is to test efficacy and safety of BAY98-7196 intravaginal ring as a new treatment option for patients with endometriosis-associated pelvic pain

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women18 years and above at the time of screening.
* Women with endometriosis confirmed by laparoscopy or laparotomy within the last ten years but not less than 8 weeks before the screening visit In Japan, diagnosis based on imaging (transvaginal ultrasound or MRI) also qualifies for inclusion.
* Moderate to severe endometriosis-associated pelvic pain (EAPP) of ≥5 in the last 28 days before screening visit 1 measured on the numeric rating scale (NRS; i.e. 4-week recall period).
* At randomization: Adherence to the study procedures during the screening period, at least 24 diary entries of ESD item 1 during the last 28 consecutive days before the randomization visit, and a sum of the available ESD item 1 ('worst pain' on the daily NRS) entries during this period of at least 98 (corresponding to an average score of ≥ 3.5).
* Willingness to use only ibuprofen as rescue pain medication for EAPP, if needed according to investigator's instruction.
* Use of a non-hormonal barrier method (i.e. spermicide-coated condoms) for contraception from screening visit until the end of the study. This is not required if adequate contraception is achieved by vasectomy of the partner

Exclusion Criteria:

* Pregnancy or lactation (less than three months since delivery, abortion, or lactation before start of treatment)
* Any diseases or conditions that can compromise the function of the body systems and could result in altered absorption, excessive accumulation, impaired metabolism, or altered excretion of the study drug
* Any diseases or conditions that might interfere with the conduct of the study or the interpretation of the results.
* Any disease or condition that may worsen under hormonal treatment according to the assessment and opinion of the investigator.
* Undiagnosed abnormal genital bleeding
* Wish for pregnancy during the study
* Regular use of pain medication due to other underlying diseases
* Non-responsiveness of endometriosis associated pelvic pain (EAPP) to GnRH-a or surgery (partial response is not exclusionary).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2014-10-16 (Actual); Primary Completion 2016-10-24 (Actual); Study Completion 2016-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (108):
- United States (25):
  - San Diego, California
  - San Francisco, California
  - Gainesville, Florida
  - New Port Richey, Florida
  - Atlanta, Georgia
  - Sandy Springs, Georgia
  - Chicago, Illinois
  - Palos Heights, Illinois
  - Wichita, Kansas
  - Marrero, Louisiana
  - Canton, Michigan
  - Detroit, Michigan
  - Saginaw, Michigan
  - Lincoln, Nebraska
  - Neptune City, New Jersey
  - Plainsboro, New Jersey
  - Durham, North Carolina
  - Greensboro, North Carolina
  - Winston-Salem, North Carolina
  - Columbus, Ohio
  - Dayton, Ohio
  - Philadelphia, Pennsylvania
  - Chattanooga, Tennessee
  - Seattle, Washington
  - Madison, Wisconsin
- Austria (4):
  - Villach, Carinthia
  - Innsbruck, Tyrol
  - Linz, Upper Austria
  - Vienna
- Belgium (3):
  - Bruxelles - Brussel
  - Edegem
  - Ghent
- Canada (5):
  - Hamilton, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec
- Czechia (8):
  - Brno
  - České Budějovice
  - Hradec Králové
  - Olomouc
  - Pilsen
  - Písek
  - Prague
  - Tábor
- Denmark (3):
  - Aarhus N
  - Copenhagen
  - Odense C
- Finland (7):
  - Espoo
  - Helsinki
  - Hyvinkää
  - Jyväskylä
  - Kuopio
  - Oulu
  - Turku
- Germany (13):
  - Karlsruhe, Baden-Wurttemberg
  - Mannheim, Baden-Wurttemberg
  - Erlangen, Bavaria
  - München, Bavaria
  - Aachen, North Rhine-Westphalia
  - Cologne, North Rhine-Westphalia
  - Dippoldiswalde, Saxony
  - Dresden, Saxony
  - Bernburg, Saxony-Anhalt
  - Blankenburg, Saxony-Anhalt
  - Jena, Thuringia
  - Berlin
  - Hamburg
- Japan (13):
  - Kitakyushu, Fukuoka
  - Sapporo, Hokkaido
  - Kawanishi, Hyōgo
  - Kanazawa, Ishikawa-ken
  - Kurashiki, Okayama-ken
  - Sayama, Osaka
  - Hamamatsu, Shizuoka
  - Bunkyo-ku, Tokyo
  - Minatoku, Tokyo
  - Shinagawa-ku, Tokyo
  - Kumamoto
  - Nagano
  - Osaka
- Netherlands (4):
  - Almere Stad
  - Groningen
  - Nieuwegein
  - Zwolle
- Norway (5):
  - Asker
  - Stokmarknes
  - Tromsø
  - Trondheim
  - Tønsberg
- Poland (7):
  - Bialystok
  - Katowice
  - Krakow
  - Lodz
  - Lublin
  - Szczecin
  - Łęczna
- Spain (7):
  - Aravaca, Madrid
  - Collado Villalba, Madrid
  - Pozuelo de Alarcón, Madrid
  - Barcelona
  - Seville
  - Valencia
  - Vitoria-Gasteiz, Álava
- Switzerland (4):
  - Lausanne, Canton of Vaud
  - Bern
  - Frauenklinik
  - Lucerne

REFERENCES:
- See also: Click here to find information about studies related to Bayer AG products conducted in Europe. — https://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted in fourteen countries in Austria, Belgium, Canada, Czech Republic, Denmark, Finland, Germany, Japan, Netherlands, Norway, Poland, Spain, Switzerland, United States, between 16 October 2014 (first participant first visit) and 24 October 2016 (last participant last visit).
Pre-assignment Details: Overall, 605 participants were screened, of them 286 failed screening, remaining 319 participants were randomized and allocated to treatment, of them 14 participants did not receive study treatment for various reasons, remaining 305 participants were treated and 272 participants completed study treatment.
Groups:
- LNG 40 mcg IVR + Placebo Injection: Participants wore an intra-vaginal ring (IVR) of Levonorgestrel (LNG) 40 microgram (mcg) continuously for 84 days, with exchange of the IVR every 28 days and participants were administered a single dose of placebo matched to leuprorelin intramuscular (i.m.) injection (3 month depot) on the first day of study treatment.
- ATZ 300 mcg / LNG 40 mcg IVR + Placebo Injection: Participants wore IVR of Anastrozole (ATZ) 300 mcg and LNG 40 mcg (BAY98-7196) continuously for 84 days, with exchange of the IVR every 28 days and participants were administered a single dose of placebo matched to leuprorelin i.m. injection (3 month depot) on the first day of study treatment.
- ATZ 600 mcg / LNG 40 mcg IVR + Placebo Injection: Participants wore IVR of ATZ 600 mcg and LNG 40 mcg (BAY98-7196) continuously for 84 days, with exchange of the IVR every 28 days and participants were administered a single dose of placebo matched to leuprorelin i.m. injection (3 month depot) on the first day of study treatment.
- ATZ 1050 mcg / LNG 40 mcg IVR + Placebo Injection: Participants wore IVR of ATZ 1050 mcg and LNG 40 mcg (BAY98-7196) continuously for 84 days, with exchange of the IVR every 28 days and participants were administered a single dose of placebo matched to leuprorelin i.m. injection (3 month depot) on the first day of study treatment.
- Placebo IVR + Leuprorelin Injection: Participants wore IVR of placebo matched to BAY98-7196 continuously for 84 days, with exchange of the IVR every 28 days and participants were administered a single dose of 11.25 milligram (mg) leuprorelin i.m. injection (3 month depot) on the first day of study treatment.
- Placebo IVR + Placebo Injection: Participants wore IVR of placebo matched to BAY98-7196 continuously for 84 days, with exchange of the IVR every 28 days and participants were administered a single dose of placebo matched to leuprorelin i.m. injection (3 month depot) on the first day of study treatment.
Period: Overall Study
Arm/Group | LNG 40 mcg IVR + Placebo Injection | ATZ 300 mcg / LNG 40 mcg IVR + Placebo Injection | ATZ 600 mcg / LNG 40 mcg IVR + Placebo Injection | ATZ 1050 mcg / LNG 40 mcg IVR + Placebo Injection | Placebo IVR + Leuprorelin Injection | Placebo IVR + Placebo Injection
Started | 52 | 53 | 55 | 53 | 53 | 53
Treated | 49 | 50 | 54 | 49 | 50 | 53
Completed | 45 | 39 | 50 | 46 | 46 | 46
Not Completed | 7 | 14 | 5 | 7 | 7 | 7
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0 | 0 | 3
Not completed — Adverse Event | 4 | 8 | 3 | 4 | 3 | 3
Not completed — Other Reasons | 1 | 2 | 0 | 2 | 0 | 0
Not completed — Lack of Efficacy | 0 | 2 | 1 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 2 | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LNG 40 mcg IVR + Placebo Injection | ATZ 300 mcg / LNG 40 mcg IVR + Placebo Injection | ATZ 600 mcg / LNG 40 mcg IVR + Placebo Injection | ATZ 1050 mcg / LNG 40 mcg IVR + Placebo Injection | Placebo IVR + Leuprorelin Injection | Placebo IVR + Placebo Injection | Total
Number analyzed (Participants) | 52 | 53 | 55 | 53 | 53 | 53 | 319
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.27 (7.4) | 32.96 (8.79) | 33.96 (5.73) | 33.72 (7.85) | 33.7 (6.29) | 34.89 (7.13) | 33.75 (7.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 53 | 55 | 53 | 53 | 53 | 319
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 24.19 (4.52) | 26.07 (6.71) | 23.84 (6.15) | 25.47 (5.68) | 25.47 (5.51) | 24.43 (5.08) | 24.91 (5.67)
Mean Pain of the 7 Days With Worst Endometriosis Associated Pelvic Pain (EAPP) [Mean (Standard Deviation); unit: units on a scale] — Pain intensity was assessed on 11-point (0-10) NRS by question 1. In question 1, participants were asked to rate the pain in the target area during the past 24 hours, where 0= no pain and 10= worst imaginable pain and responses were recorded in ESD. The mean pain of the 7 days with worst EAPP within a 28-day window was calculated as the sum of ESD item 1 on 7 days with worst EAPP within that 28-day window divided by 7.
  units on a scale | 7.8205 (1.171) | 7.4664 (0.9893) | 8.1905 (1.068) | 7.5429 (1.2568) | 7.8964 (1.1952) | 7.6886 (1.2389) | 7.7842 (1.1702)
Percentage of Days With Pain Greater Than or Equal to (>=) 7 [Mean (Standard Deviation); unit: percentage of days] — Higher numbers are associated with more days of pain above the 7 on the 11-point (0-10) NRS.
  percentage of days | 50.094 (35.5201) | 40.1521 (29.8714) | 55.1155 (33.7625) | 37.3044 (30.2894) | 48.7001 (33.6685) | 41.1847 (33.0479) | 45.8234 (33.1247)
Percentage of Days With Pain >=4 [Mean (Standard Deviation); unit: percentage of days] — Higher numbers are associated with more days of pain above the 4 on the 11-point (0-10) NRS.
  percentage of days | 86.0058 (19.3136) | 84.7239 (18.1713) | 89.029 (16.3667) | 85.8451 (17.9466) | 92.9141 (11.6008) | 80.4397 (20.1004) | 86.6042 (17.6568)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Mean Pain of the 7 Days With Worst EAPP From Baseline (Last 28 Days Before Randomization) to End of Treatment (Last 28 Days of Treatment Period, Days 57-84) as Measured on NRS by Question 1 of ESD
Description: Pain intensity was assessed on 11-point (0-10) NRS by question 1. In question 1, participants were asked to rate the pain in the target area during the past 24 hours, where 0= no pain and 10= worst imaginable pain and responses were recorded in ESD. The mean pain of the 7 days with worst EAPP within a 28-day window was calculated as the sum of ESD item 1 on 7 days with worst EAPP within that 28-day window divided by 7.
Time Frame: Baseline (last 28 days before randomization), end of treatment (Treatment 3) (last 28 days of the treatment period, Day 57-84)
Population: The dose-response analysis was performed using the MCP-Mod method with groups containing LNG, ATZ + LNG, and Placebo. It was analyzed using the per-protocol set (PPS) with evaluable participants for this endpoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LNG 40 mcg IVR + Placebo Injection | ATZ 300 mcg / LNG 40 mcg IVR + Placebo Injection | ATZ 600 mcg / LNG 40 mcg IVR + Placebo Injection | ATZ 1050 mcg / LNG 40 mcg IVR + Placebo Injection | Placebo IVR + Leuprorelin Injection | Placebo IVR + Placebo Injection
Number analyzed (Participants) | 39 | 33 | 42 | 35 | 40 | 39
units on a scale | -1.8974 (1.6416) [lower limit 1.6416] | -1.6061 (1.6652) [lower limit 1.6652] | -2.4014 (2.1833) [lower limit 2.1833] | -2.2653 (1.5972) [lower limit 1.5972] | -3.7679 (2.3507) [lower limit 1.8247] | -2.293 (1.8247)
Statistical Analysis 1: Comparison: LNG 40 mcg IVR + Placebo Injection vs ATZ 300 mcg / LNG 40 mcg IVR + Placebo Injection vs ATZ 600 mcg / LNG 40 mcg IVR + Placebo Injection vs ATZ 1050 mcg / LNG 40 mcg IVR + Placebo Injection vs Placebo IVR + Leuprorelin Injection; The analysis was performed by using MCP-Mod method using pre-defined candidate dose-response model; Test type: Superiority or Other; p = 0.3875, Contrast tests for dose-response model; Emax = 0.1483, Standard Error of Mean 0.2925
Statistical Analysis 2: Comparison: LNG 40 mcg IVR + Placebo Injection vs ATZ 300 mcg / LNG 40 mcg IVR + Placebo Injection vs ATZ 600 mcg / LNG 40 mcg IVR + Placebo Injection vs ATZ 1050 mcg / LNG 40 mcg IVR + Placebo Injection vs Placebo IVR + Leuprorelin Injection; The analysis was performed by using MCP-Mod method using pre-defined candidate dose-response model; Test type: Superiority or Other; p = 0.2676, Contrast tests for dose-response model; Linear = 0.2484, Standard Error of Mean 0.2975
Statistical Analysis 3: Comparison: LNG 40 mcg IVR + Placebo Injection vs ATZ 300 mcg / LNG 40 mcg IVR + Placebo Injection vs ATZ 600 mcg / LNG 40 mcg IVR + Placebo Injection vs ATZ 1050 mcg / LNG 40 mcg IVR + Placebo Injection vs Placebo IVR + Leuprorelin Injection; The analysis was performed by using MCP-Mod method using pre-defined candidate dose-response model; Test type: Superiority or Other; p = 0.3211, Contrast tests for dose-response model; Sigmoidal Emax 1 = 0.1995, Standard Error of Mean 0.2922
Statistical Analysis 4: Comparison: LNG 40 mcg IVR + Placebo Injection vs ATZ 300 mcg / LNG 40 mcg IVR + Placebo Injection vs ATZ 600 mcg / LNG 40 mcg IVR + Placebo Injection vs ATZ 1050 mcg / LNG 40 mcg IVR + Placebo Injection vs Placebo IVR + Leuprorelin Injection; The analysis was performed by using MCP-Mod method using pre-defined candidate dose-response model; Test type: Superiority or Other; p = 0.1721, Contrast tests for dose-response model; Sigmoidal Emax 2 = 0.3467, Standard Error of Mean 0.2994

2. Secondary Outcome: Absolute Change in Mean Pain of the 7 Days With Worst EAPP From Baseline (Last 28 Days Before Randomization) to First Cycle Under Study Treatment (Day 1-28) and to Second Cycle Under Study Treatment (Day 29-56) as Measured on NRS by Question 1 of ESD
Description: Pain intensity was assessed on 11-point (0-10) NRS by question 1. In question 1, subjects were asked to rate the pain in the target area during the past 24 hours, where 0= no pain and 10= worst imaginable pain and responses were recorded in ESD. The mean pain of the 7 days with worst EAPP within a 28-day window was calculated as the sum of ESD item 1 on 7 days with worst EAPP within that 28-day window divided by 7.
Time Frame: Baseline (last 28 days before randomization), first cycle (Treatment 1) (Day 1-28), second cycle (Treatment 2) (Day 29-56)
Population: It was analyzed using the per-protocol set (PPS) with evaluable participants for this endpoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LNG 40 mcg IVR + Placebo Injection | ATZ 300 mcg / LNG 40 mcg IVR + Placebo Injection | ATZ 600 mcg / LNG 40 mcg IVR + Placebo Injection | ATZ 1050 mcg / LNG 40 mcg IVR + Placebo Injection | Placebo IVR + Leuprorelin Injection | Placebo IVR + Placebo Injection
Number analyzed (Participants) | 39 | 34 | 42 | 35 | 40 | 39
units on a scale
  Change at Treatment 1 | -0.7582 (1.1518) [lower limit 1.1518] | -0.6849 (1.3832) [lower limit 1.3832] | -1.1463 (1.3992) [lower limit 1.3992] | -1.0000 (1.2579) [lower limit 1.2579] | -1.2071 (1.1978) [lower limit 1.1978] | -0.9048 (1.1686) [lower limit 1.1686]
  Change at Treatment 2 | -1.6447 (1.4831) [lower limit 1.4831] | -1.5126 (2.0161) [lower limit 2.0161] | -2.1224 (2.2791) [lower limit 2.2791] | -1.9959 (1.3978) [lower limit 1.3978] | -2.8607 (2.0665) [lower limit 2.0665] | -1.8022 (1.5131) [lower limit 1.5131]
Statistical Analysis 1: Comparison: LNG 40 mcg IVR + Placebo Injection vs ATZ 300 mcg / LNG 40 mcg IVR + Placebo Injection vs ATZ 600 mcg / LNG 40 mcg IVR + Placebo Injection vs ATZ 1050 mcg / LNG 40 mcg IVR + Placebo Injection vs Placebo IVR + Placebo Injection; The analysis was performed by using MCP-Mod method using pre-defined candidate dose-response model; Test type: Superiority or Other; p = 0.231, Contrast tests for dose-response model; Emax = 0.2736, Standard Error of Mean 0.2878
Statistical Analysis 2: Comparison: LNG 40 mcg IVR + Placebo Injection vs ATZ 300 mcg / LNG 40 mcg IVR + Placebo Injection vs ATZ 600 mcg / LNG 40 mcg IVR + Placebo Injection vs ATZ 1050 mcg / LNG 40 mcg IVR + Placebo Injection vs Placebo IVR + Placebo Injection; The analysis was performed by using MCP-Mod method using pre-defined candidate dose-response model; Test type: Superiority or Other; p = 0.1865, Contrast tests for dose-response model; Linear = 0.3234, Standard Error of Mean 0.2927
Statistical Analysis 3: Comparison: LNG 40 mcg IVR + Placebo Injection vs ATZ 300 mcg / LNG 40 mcg IVR + Placebo Injection vs ATZ 600 mcg / LNG 40 mcg IVR + Placebo Injection vs ATZ 1050 mcg / LNG 40 mcg IVR + Placebo Injection vs Placebo IVR + Placebo Injection; The analysis was performed by using MCP-Mod method using pre-defined candidate dose-response model; Test type: Superiority or Other; p = 0.1955, Contrast tests for dose-response model; Sigmoidal Emax 1 = 0.3081, Standard Error of Mean 0.2875
Statistical Analysis 4: Comparison: LNG 40 mcg IVR + Placebo Injection vs ATZ 300 mcg / LNG 40 mcg IVR + Placebo Injection vs ATZ 600 mcg / LNG 40 mcg IVR + Placebo Injection vs ATZ 1050 mcg / LNG 40 mcg IVR + Placebo Injection vs Placebo IVR + Placebo Injection; The analysis was performed by using MCP-Mod method using pre-defined candidate dose-response model; Test type: Superiority or Other; p = 0.1416, Contrast tests for dose-response model; Sigmoidal Emax 2 = 0.3781, Standard Error of Mean 0.2944

3. Secondary Outcome: Absolute Change in Mean Pain From Baseline (Last 28 Days Before Randomization) to First Cycle Under Study Treatment(Day1-28), Second Cycle Under Study Treatment(Day29-56),Third Cycle Under Study Treatment (Day57-84) as Measured on NRS by Question1 of ESD
Description: Pain intensity was assessed on 11-point (0-10) NRS by question 1. In question 1, subjects were asked to rate the pain in the target area during the past 24 hours, where 0= no pain and 10= worst imaginable pain and responses were recorded in ESD. The mean pain within a 28-day window was calculated as the sum of ESD item 1 within that 28-day window divided by the number with non-missing days within that 28-day window. Here, number of subjects 'n' signifies evaluable subjects for the respective category.
Time Frame: Baseline (last 28 days before randomization), first cycle (Treatment 1) (Day 1-28), second cycle (Treatment 2) (Day 29-56), and third cycle (Treatment 3) (last 28 days of the treatment period, Day 57-84)
Population: It was analyzed using the per-protocol set (PPS) with evaluable participants for this endpoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LNG 40 mcg IVR + Placebo Injection | ATZ 300 mcg / LNG 40 mcg IVR + Placebo Injection | ATZ 600 mcg / LNG 40 mcg IVR + Placebo Injection | ATZ 1050 mcg / LNG 40 mcg IVR + Placebo Injection | Placebo IVR + Leuprorelin Injection | Placebo IVR + Placebo Injection
Number analyzed (Participants) | 39 | 34 | 42 | 35 | 40 | 39
units on a scale
  Baseline | 6.0938 (1.5314) | 5.7409 (1.3044) | 6.3694 (1.5300) | 5.7128 (1.4415) | 6.3962 (1.4575) | 5.6399 (1.5312)
  Change at Treatment 1 | -0.8472 (1.1905) | -0.9009 (1.3434) | -1.0931 (1.4002) | -1.1257 (1.3317) | -1.5315 (1.4809) | -0.9777 (1.0680)
  Change at Treatment 2 | -1.5774 (1.6278) | -1.5068 (1.8707) | -1.7349 (1.9403) | -1.9615 (1.3966) | -2.6855 (2.0601) | -1.8994 (1.3069)
  Change at Treatment 3: number analyzed (Participants) | 39 | 33 | 42 | 35 | 40 | 39
  Change at Treatment 3 | -1.8001 (1.7687) | -1.6411 (1.8071) | -2.0112 (1.9575) | -2.1268 (1.6877) | -3.502 (2.3096) | -2.2228 (1.4957)
Statistical Analysis 1: Comparison: LNG 40 mcg IVR + Placebo Injection vs ATZ 300 mcg / LNG 40 mcg IVR + Placebo Injection vs ATZ 600 mcg / LNG 40 mcg IVR + Placebo Injection vs ATZ 1050 mcg / LNG 40 mcg IVR + Placebo Injection vs Placebo IVR + Placebo Injection; The analysis was performed by using MCP-Mod method using pre-defined candidate dose-response model; Test type: Superiority or Other; p = 0.5794, Contrast tests for dose-response model; Emax = 0.0081, Standard Error of Mean 0.2832
Statistical Analysis 2: Comparison: LNG 40 mcg IVR + Placebo Injection vs ATZ 300 mcg / LNG 40 mcg IVR + Placebo Injection vs ATZ 600 mcg / LNG 40 mcg IVR + Placebo Injection vs ATZ 1050 mcg / LNG 40 mcg IVR + Placebo Injection vs Placebo IVR + Placebo Injection; The analysis was performed by using MCP-Mod method using pre-defined candidate dose-response model; Test type: Superiority or Other; p = 0.4301, Contrast tests for dose-response model; Linear = 0.1148, Standard Error of Mean 0.2880
Statistical Analysis 3: Comparison: LNG 40 mcg IVR + Placebo Injection vs ATZ 300 mcg / LNG 40 mcg IVR + Placebo Injection vs ATZ 600 mcg / LNG 40 mcg IVR + Placebo Injection vs ATZ 1050 mcg / LNG 40 mcg IVR + Placebo Injection vs Placebo IVR + Placebo Injection; The analysis was performed by using MCP-Mod method using pre-defined candidate dose-response model; Test type: Superiority or Other; p = 0.5337, Contrast tests for dose-response model; Sigmoidal Emax 1 = 0.0401, Standard Error of Mean 0.2829
Statistical Analysis 4: Comparison: LNG 40 mcg IVR + Placebo Injection vs ATZ 300 mcg / LNG 40 mcg IVR + Placebo Injection vs ATZ 600 mcg / LNG 40 mcg IVR + Placebo Injection vs ATZ 1050 mcg / LNG 40 mcg IVR + Placebo Injection vs Placebo IVR + Placebo Injection; The analysis was performed by using MCP-Mod method using pre-defined candidate dose-response model; Test type: Superiority or Other; p = 0.3396, Contrast tests for dose-response model; Sigmoidal Emax 2 = 0.1835, Standard Error of Mean 0.2899

4. Secondary Outcome: Percentage of Days During Baseline (Last 28 Days Before Randomization) and Cycles 1, 2, and 3 With Pain Greater Than or Equal to (>=) 7 as Measured on NRS by Question 1 of ESD as Measured on NRS by Question 1 of ESD
Description: Pain intensity was assessed on 11-point (0-10) NRS by question 1. In question 1, subjects were asked to rate the pain in the target area during the past 24 hours, where 0= no pain and 10= worst imaginable pain and responses were recorded in ESD. The percentage of days with pain >=7 within a 28-day window was calculated as 100 divided by the number of non-missing days within that 28-day window multiplied by the number of days within that 28-day window where item 1 of the ESD was >=7.
Time Frame: Baseline (last 28 days before randomization), Cycle 1 (Treatment 1), Cycle 2 (Treatment 2), and Cycle 3 (Treatment 3)
Population: It was analyzed using the per-protocol set (PPS) with evaluable participants for this endpoint.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | LNG 40 mcg IVR + Placebo Injection | ATZ 300 mcg / LNG 40 mcg IVR + Placebo Injection | ATZ 600 mcg / LNG 40 mcg IVR + Placebo Injection | ATZ 1050 mcg / LNG 40 mcg IVR + Placebo Injection | Placebo IVR + Leuprorelin Injection | Placebo IVR + Placebo Injection
Number analyzed (Participants) | 41 | 34 | 42 | 35 | 41 | 39
percentage of days
  Treatment 1 | 35.6034 (34.3126) | 27.5659 (27.6426) | 40.0813 (37.2694) | 23.9322 (28.6234) | 28.2015 (28.8430) | 25.1742 (24.2811)
  Treatment 2 | 25.6257 (33.9315) | 22.8695 (28.3443) | 34.4364 (40.5623) | 14.9331 (23.8028) | 12.1320 (25.1638) | 14.1869 (17.7364)
  Treatment 3: number analyzed (Participants) | 41 | 33 | 42 | 35 | 41 | 39
  Treatment 3 | 23.1293 (33.9451) | 19.9332 (26.0540) | 29.8103 (39.0434) | 14.3362 (25.6770) | 8.5351 (20.7819) | 12.7574 (18.5154)

5. Secondary Outcome: Change From Baseline (Last 28 Days Before Randomization) to Cycle 1, 2, and 3 in Percentage of Days With Pain >=7 as Measured on NRS by Question 1 of ESD
Description: Pain intensity was assessed on 11-point (0-10) NRS by question 1. In question 1, subjects were asked to rate the pain in the target area during the past 24 hours, where 0= no pain and 10= worst imaginable pain and responses were recorded in ESD. The percentage of days with pain >=7 within a 28-day window was calculated as 100 divided by the number of non-missing days within that 28-day window multiplied by the number of days within that 28-day window where item 1 of the ESD was >=7. Here, number of subjects 'n' signifies evaluable subjects for the respective category.
Time Frame: Baseline (last 28 days before randomization), Cycle 1 (Treatment 1), Cycle 2 (Treatment 2), and Cycle 3 (Treatment 3)
Population: It was analyzed using the per-protocol set (PPS) with evaluable participants for this endpoint.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | LNG 40 mcg IVR + Placebo Injection | ATZ 300 mcg / LNG 40 mcg IVR + Placebo Injection | ATZ 600 mcg / LNG 40 mcg IVR + Placebo Injection | ATZ 1050 mcg / LNG 40 mcg IVR + Placebo Injection | Placebo IVR + Leuprorelin Injection | Placebo IVR + Placebo Injection
Number analyzed (Participants) | 39 | 34 | 42 | 35 | 40 | 39
percentage of days
  Change at Treatment 1 | -13.6756 (22.6822) | -12.5862 (21.4336) | -15.0341 (21.0071) | -13.3722 (19.6416) | -19.8898 (25.9273) | -16.0105 (19.0190)
  Change at Treatment 2 | -24.1404 (28.5082) | -17.2826 (29.0007) | -20.6791 (30.2152) | -22.3713 (24.4098) | -36.3540 (34.9706) | -26.9979 (24.9493)
  Change at Treatment 3: number analyzed (Participants) | 39 | 33 | 42 | 35 | 40 | 39
  Change at Treatment 3 | -26.4197 (31.4648) | -20.8529 (28.3939) | -25.3052 (33.5497) | -22.9682 (28.8677) | -39.9516 (33.8277) | -28.4273 (29.6186)

6. Secondary Outcome: Percentage of Days During Baseline (Last 28 Days Before Randomization) and Cycles 1, 2, and 3 With Pain >=4 as Measured on NRS by Question 1 of ESD
Description: Pain intensity was assessed on 11-point (0-10) NRS by question 1. In question 1, subjects were asked to rate the pain in the target area during the past 24 hours, where 0= no pain and 10= worst imaginable pain and responses were recorded in ESD. The percentage of days with pain >=4 within a 28-day window was calculated as 100 divided by the number of non-missing days within that 28-day window multiplied by the number of days within that window where Item 1 of the ESD was >=4. Here, number of subjects 'n' signifies evaluable subjects for the respective category.
Time Frame: Baseline (last 28 days before randomization), Cycle 1 (Treatment 1), Cycle 2 (Treatment 2), and Cycle 3 (Treatment 3)
Population: It was analyzed using the per-protocol set (PPS) with evaluable participants for this endpoint.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | LNG 40 mcg IVR + Placebo Injection | ATZ 300 mcg / LNG 40 mcg IVR + Placebo Injection | ATZ 600 mcg / LNG 40 mcg IVR + Placebo Injection | ATZ 1050 mcg / LNG 40 mcg IVR + Placebo Injection | Placebo IVR + Leuprorelin Injection | Placebo IVR + Placebo Injection
Number analyzed (Participants) | 41 | 34 | 42 | 35 | 41 | 39
percentage of days
  Treatment 1 | 71.8037 (32.3658) | 69.3092 (27.8642) | 73.8956 (31.6868) | 70.6504 (27.8528) | 70.2066 (28.9333) | 65.9074 (30.0166)
  Treatment 2 | 61.8199 (37.1217) | 57.8777 (34.7429) | 62.5822 (37.6989) | 52.6028 (35.6106) | 54.0965 (38.9629) | 49.487 (31.3566)
  Treatment 3: number analyzed (Participants) | 41 | 33 | 42 | 35 | 41 | 39
  Treatment 3 | 60.2902 (37.8585) | 57.0171 (34.3642) | 56.7691 (40.3803) | 50.7332 (36.2903) | 38.6986 (39.6045) | 47.0976 (35.3227)

7. Secondary Outcome: Change From Baseline (Last 28 Days Before Randomization) to Cycle 1, 2, and 3 in Percentage of Days With Pain >=4 as Measured on NRS by Question 1 of ESD
Description: as for outcome 6
Time Frame: Baseline (last 28 days before randomization), Cycle 1 (Treatment 1), Cycle 2 (Treatment 2), and Cycle 3 (Treatment 3)
Population: It was analyzed using the per-protocol set (PPS) with evaluable participants for this endpoint.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | LNG 40 mcg IVR + Placebo Injection | ATZ 300 mcg / LNG 40 mcg IVR + Placebo Injection | ATZ 600 mcg / LNG 40 mcg IVR + Placebo Injection | ATZ 1050 mcg / LNG 40 mcg IVR + Placebo Injection | Placebo IVR + Leuprorelin Injection | Placebo IVR + Placebo Injection
Number analyzed (Participants) | 39 | 34 | 42 | 35 | 40 | 39
percentage of days
  Change at Treatment 1 | -12.8228 (20.4330) | -15.4147 (24.0608) | -15.1334 (22.5347) | -15.1947 (21.1740) | -21.4331 (23.4546) | -14.5323 (20.9670)
  Change at Treatment 2 | -22.4950 (28.1535) | -26.8462 (32.6194) | -26.4468 (34.4661) | -33.2423 (27.3686) | -37.7330 (36.9484) | -30.9527 (25.4665)
  Change at Treatment 3: number analyzed (Participants) | 39 | 33 | 42 | 35 | 40 | 39
  Change at Treatment 3 | -23.5498 (30.2853) | -27.4770 (34.2051) | -32.2600 (37.4997) | -35.1119 (30.9316) | -53.4266 (38.8452) | -33.3421 (25.7105)

ADVERSE EVENTS:
Time Frame: From start of study treatment up to 30 days after end of treatment (Day 114)
Arm/Group | LNG 40 mcg IVR + Placebo Injection | ATZ 300 mcg / LNG 40 mcg IVR + Placebo Injection | ATZ 600 mcg / LNG 40 mcg IVR + Placebo Injection | ATZ 1050 mcg / LNG 40 mcg IVR + Placebo Injection | Placebo IVR + Leuprorelin Injection | Placebo IVR + Placebo Injection
Serious Adverse Events (participants affected / at risk) | 2/49 | 0/50 | 0/54 | 2/49 | 3/50 | 4/53
Other Adverse Events (participants affected / at risk) | 38/49 | 40/50 | 40/54 | 35/49 | 35/50 | 38/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LNG 40 mcg IVR + Placebo Injection (N=49) | ATZ 300 mcg / LNG 40 mcg IVR + Placebo Injection (N=50) | ATZ 600 mcg / LNG 40 mcg IVR + Placebo Injection (N=54) | ATZ 1050 mcg / LNG 40 mcg IVR + Placebo Injection (N=49) | Placebo IVR + Leuprorelin Injection (N=50) | Placebo IVR + Placebo Injection (N=53)
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pregnancy of unknown location (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Renal atrophy (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 1 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LNG 40 mcg IVR + Placebo Injection (N=49) | ATZ 300 mcg / LNG 40 mcg IVR + Placebo Injection (N=50) | ATZ 600 mcg / LNG 40 mcg IVR + Placebo Injection (N=54) | ATZ 1050 mcg / LNG 40 mcg IVR + Placebo Injection (N=49) | Placebo IVR + Leuprorelin Injection (N=50) | Placebo IVR + Placebo Injection (N=53)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 1
Haemorrhagic disorder (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Deafness transitory (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 1 | 0
Conjunctivitis allergic (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Eyelid rash (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 4 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 0 | 3 | 1 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 2 | 2 | 4 | 3 | 3
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Dyschezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Noninfectious peritonitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Faeces soft (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 1 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 3 | 1 | 1 | 0 | 2
Feeling hot (General disorders) | 0 | 0 | 1 | 1 | 0 | 0
Hunger (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Injection site reaction (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 1 | 0
Pelvic mass (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 0 | 0 | 0 | 0
Swelling (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Peripheral swelling (General disorders) | 0 | 1 | 1 | 0 | 1 | 0
Medical device discomfort (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhagic cyst (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Medical device site discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 2
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bacterial vaginosis (Infections and infestations) | 1 | 0 | 2 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 1 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 2 | 1 | 2 | 1 | 0 | 1
Ear infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 2 | 1 | 2 | 0
Hordeolum (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 2 | 0 | 1 | 3 | 0
Nasopharyngitis (Infections and infestations) | 2 | 2 | 7 | 5 | 1 | 3
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pulpitis dental (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 1 | 2 | 0
Tonsillitis (Infections and infestations) | 1 | 1 | 3 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0
Urethritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 2 | 2 | 1 | 1 | 2
Vulvovaginal candidiasis (Infections and infestations) | 2 | 0 | 0 | 1 | 0 | 0
Nail infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Borrelia infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 2 | 1 | 2 | 1 | 2 | 2
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Bone contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Closed globe injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0 | 1 | 0 | 0
Alanine aminotransferase abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 2 | 0 | 0 | 0 | 1
Aspartate aminotransferase abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Colonoscopy (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Blood urine present (Investigations) | 1 | 1 | 0 | 0 | 0 | 0
Prothrombin time shortened (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Red blood cells urine positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Weight increased (Investigations) | 2 | 1 | 1 | 1 | 0 | 1
White blood cells urine positive (Investigations) | 3 | 1 | 0 | 0 | 0 | 0
Urine bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Nitrite urine present (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
Protein urine present (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Urine ketone body present (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Smear vaginal abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Gardnerella test positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 1 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 0 | 2 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 2 | 3
Headache (Nervous system disorders) | 5 | 8 | 3 | 8 | 8 | 6
Migraine (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 2 | 1 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 2 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 2 | 0
Irritability (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Libido decreased (Psychiatric disorders) | 0 | 1 | 1 | 0 | 4 | 0
Loss of libido (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 1 | 1 | 1 | 0
Mood swings (Psychiatric disorders) | 1 | 1 | 2 | 0 | 0 | 2
Depressive symptom (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Affect lability (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1
Amenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Breast cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Breast enlargement (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 2 | 2 | 1 | 0 | 2 | 0
Breast tenderness (Reproductive system and breast disorders) | 0 | 1 | 1 | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1 | 2
Dyspareunia (Reproductive system and breast disorders) | 1 | 1 | 0 | 0 | 3 | 0
Endometriosis (Reproductive system and breast disorders) | 3 | 2 | 3 | 2 | 2 | 5
Fibrocystic breast disease (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 1
Galactorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hydrosalpinx (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypomenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 1 | 1 | 1 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 2
Metrorrhagia (Reproductive system and breast disorders) | 1 | 1 | 2 | 2 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 20 | 20 | 24 | 16 | 5 | 7
Ovarian rupture (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 1 | 2 | 2 | 0 | 2
Polymenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 0 | 2 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 3 | 2 | 4 | 0 | 0
Vaginal odour (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Varicose veins pelvic (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 4 | 1
Breast discomfort (Reproductive system and breast disorders) | 0 | 1 | 1 | 1 | 0 | 0
Adenomyosis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 0 | 1
Adnexa uteri pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 1
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0 | 2 | 0 | 2 | 0 | 0
Genital haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 1 | 1 | 1 | 0
Uterine haematoma (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vaginal flatulence (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vulvovaginal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abnormal withdrawal bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 5 | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hand dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Wisdom teeth removal (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 3 | 3 | 17 | 2
Device breakage (Product Issues) | 0 | 0 | 0 | 0 | 0 | 1
Device expulsion (Product Issues) | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a period of five (5) years from the date of last disclosure under this Agreement. Recipient shall (a) maintain all Confidential Information in confidence and not disclose the same to any third party unless required to do so by court order or by law, in which case Recipient shall notify Bayer in writing prior to making such a disclosure, and (b) not use any Confidential Information for its own benefit or for the benefit of any third party.